CLINICAL TRIAL: NCT01374854
Title: Umbilical Mesenchymal Stem Cells and Mononuclear Cells Infusion in Type 1 Diabetes Mellitus: A Randomized Controlled Open-label Study
Brief Title: Umbilical Mesenchymal Stem Cells and Mononuclear Cells Infusion in Type 1 Diabetes Mellitus
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCMSC-T1DM
Record Dates: First submitted 2011-06-15; First posted 2011-06-16 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: type 1 diabetes mellitus; umbilical mesenchymal stem cell; mononuclear cell
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stem Cell Infusion (Experimental)
  Interventions: Biological: Umbilical mesenchymal stem cell (UC-MSCs) infusion
- traditional therapy control (Active Comparator)
  Interventions: Drug: traditional therapy

INTERVENTIONS:
Biological: Umbilical mesenchymal stem cell (UC-MSCs) infusion — 1×10^6/kg UC-MSCs is infused through pancreatic artery along with mononuclear cells by interventional therapy and another same dose of UC-MSCs is administered one week post-intervention.
  Arms: Stem Cell Infusion
Drug: traditional therapy — exogenous insulin injection daily
  Arms: traditional therapy control

SUMMARY:
Umbilical mesenchymal stem cells (UC-MSCs) infusion is supposed be a promising regeneration therapy with mild side effect as indicated by large quantities of animal experiments and some clinical trials. There are few UC-MSCs clinical trials with regard to diabetes mellitus. The investigators hypothesize that infusion of USC-MSCs may provide multiple signals for beta-cell regeneration and even re-differentiate into local tissues in diabetes mellitus patients, resulting in improvement of diabetic control, of which the effect may be promoted by concomitant infusion of bone marrow mononuclear cells and maximized by intra-arterial pancreatic infusion through angiography.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age 18 to 65 years of age.
* Ability to provide written informed consent.
* Mentally stable and able to comply with the procedures of the study protocol.
* Clinical history compatible with type 1 diabetes (T1DM) as defined by the Expert Committee on the Diagnosis and classification of Diabetes Mellitus
* Onset of T1DM disease at ≤ 35 years of age.
* T1DM duration ≥ 2 and ≤ 20 years at the time of enrollment.
* Basal C-peptide ≤ 0.3 ng/mL
* HbA1c ≥ 7.5 at time of enrollment.

Exclusion Criteria:

* BMI >35 kg/m^2.
* Insulin requirements of > 100 U/day.
* C-reactive protein (hs-CRP) >3.00ng/ml
* Uncontrolled blood Pressure: SBP >160 mmHg or DBP >100 mmHg at the time of enrollment.
* Evidence of renal dysfunction, serum creatinine > 1.5 mg/dl (males) and 1.4 mg/dl (females).
* Proteinuria > 300 mg/day
* Evidence of cardiovascular disease, existing congestive cardiac failure on physical exam and/or acute coronary syndrome in past 6 months.
* For female participants: Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study. For male participants: intent to procreate 3 months before or after the intervention or unwillingness to use effective measures of contraception. Oral contraceptives, Norplant®, Depo-Provera®, and barrier devices with spermicide are acceptable contraceptive methods; condoms used alone are not acceptable
* Active infection including hepatitis C, HIV, or TB as determined by a positive skin test or clinical presentation, or under treatment for suspected TB. Positive tests are acceptable only if associated with a history of previous vaccination in the absence of any sign of active infection. Positive tests are otherwise not acceptable, even in the absence of any active infection at the time of evaluation
* Known active alcohol or substance abuse including cigarette/cigar smoking
* Baseline Hemoglobin below the lower limits of normal at the local laboratory; lymphopenia (<1,000/L), neutropenia (<1,500/L), or thrombocytopenia (platelets <100,000/L).
* A history of Factor V deficiency or other coagulopathy defined by INR >1.5, PTT >40, PT >15.
* Any coagulopathy or medical condition requiring long-term anticoagulant therapy (e.g., warfarin) after transplantation (low-dose aspirin treatment is allowed) or patients with an INR >1.5.
* Acute or chronic pancreatitis.
* Symptomatic peptic ulcer disease.
* Hyperlipidemia despite medical therapy (fasting LDL cholesterol >130 mg/dl, treated or untreated; and/or fasting triglycerides > 200 mg/dl).
* Receiving treatment for a medical condition requiring chronic use of systemic steroids.
* Symptomatic cholecystolithiasis.
* Use of any investigational agents within 4 weeks of enrollment.
* Admission to hospital for any reason in the 14 days prior to enrollment (signing consent).
* Presence of active proliferative diabetic retinopathy or macular edema
* Any malignancy
* Abnormal liver function >1.5 x ULN
* Abdominal aortic aneurysm
* History of cerebro-vascular accident
* Any patient with acute or subacute decompensation from diabetes
* Any acute or chronic infectious condition that in the criteria of the investigator would be a risk for the patient.
* Subjects with hypoproteinemia, cachexia or terminal states
* Subjects with history of anorexia/bulimia
* Subjects with respiratory insufficiency
* Any medical condition that, in the opinion of the investigator, will interfere with the safe completion of the trial.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
c-peptide area under the curve during OGTT | 1 year

SECONDARY OUTCOMES:
The incidence and severity of adverse events related to the stem cell infusion procedure | 1 year
The reduction in fasting blood glucose (FBG) | 1 year
The increase in basal C-peptide | 1 year
The reduction in exogenous insulin requirements | 1 year
Decrease in HbA1c | 1 year
insulin area under the curve during OGTT | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Tan, professor, Principal Investigator — Fuzhou General Hospital
Locations (1):
- Fuzhou General Hospital, Fuzhou, Fujian, China

REFERENCES:
- [Derived] Wu Z, Xu X, Cai J, Chen J, Huang L, Wu W, Pugliese A, Li S, Ricordi C, Tan J. Prevention of chronic diabetic complications in type 1 diabetes by co-transplantation of umbilical cord mesenchymal stromal cells and autologous bone marrow: a pilot randomized controlled open-label clinical study with 8-year follow-up. Cytotherapy. 2022 Apr;24(4):421-427. doi: 10.1016/j.jcyt.2021.09.015. Epub 2022 Jan 25. PMID 35086778
- [Derived] Cai J, Wu Z, Xu X, Liao L, Chen J, Huang L, Wu W, Luo F, Wu C, Pugliese A, Pileggi A, Ricordi C, Tan J. Umbilical Cord Mesenchymal Stromal Cell With Autologous Bone Marrow Cell Transplantation in Established Type 1 Diabetes: A Pilot Randomized Controlled Open-Label Clinical Study to Assess Safety and Impact on Insulin Secretion. Diabetes Care. 2016 Jan;39(1):149-57. doi: 10.2337/dc15-0171. Epub 2015 Dec 1. PMID 26628416